CLINICAL TRIAL: NCT04713657
Title: Mechanistic Clinical Trial of Beta-Blocker Administration For Reactivating Cardiomyocyte Division In Tetralogy of Fallot
Brief Title: Beta-blocker Administration for Cardiomyocyte Division
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-12026881; R01HL155597 (NIH)
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Tetralogy of Fallot; Double Outlet Right Ventricle
Keywords: Tetralogy of Fallot; Double Outlet Right Ventricle
MeSH Terms: conditions — Tetralogy of Fallot; Double Outlet Right Ventricle | interventions — Thymidine; Urine Specimen Collection; Propranolol; Restraint, Physical; Specimen Handling

STUDY DESIGN:
Intervention Model Description: double-blinded, placebo-controlled (1:1) randomized, single-center trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propranolol (Active Comparator): The target dose of Propranolol hydrochloride for this study target dose for this study will be 4 mg/kg/day divided in 4 doses. The concentration of propranolol solution is 20 mg/5 mL. Additionally, labeled syringes will be provided to families for accurate weight-based dosing. Treatment with propranolol will begin at 1 month of age and continue until 4 months of age or 24hrs prior to surgical repair, whichever comes first.
  Interventions: Other: N-thymidine; Other: Urine Collection; Procedure: Echocardiogram; Procedure: Cardiac MRI (CMR); Drug: Propranolol Hydrochloride; Procedure: Physical Exam; Other: Specimen Collection
- Placebo (Placebo Comparator): Placebo will be given in a volume that corresponds to the patient's weight. Additionally, labeled syringes will be provided to families for accurate weight-based dosing. Treatment with placebo will begin at 1 month of age and continue until 4 months of age or 24hrs prior to surgical repair, whichever comes first. There is no current standard of care for pharmacologic therapy for infants with Tetralogy of Fallot (ToF). As such, there are no alternative treatments, and the placebo group is standard of care.
  Interventions: Other: N-thymidine; Other: Urine Collection; Procedure: Echocardiogram; Procedure: Cardiac MRI (CMR); Drug: Placebo; Procedure: Physical Exam; Other: Specimen Collection

INTERVENTIONS:
Other: N-thymidine — 15N-thymidine will be administered to patients in order to quantify cardiomyocyte proliferation. 15N-thymidine will be administered as 5 separate syringes. Each syringe will contain the recommended daily dose based on participants weight. Subjects will be given the labeled thymidine by mouth once a day for 5 consecutive days. The dosing will begin one week after starting the study drug.The caregiver (parent or nurse) will administer the labeled thymidine by mouth via a syringe once a day for 5 consecutive days. They will be provided with a diary to keep track of study drug dosing.
  Other Names: Thymidine
Other: Urine Collection — Parents will be asked to keep a diary of the child's feeding and diaper changes during the administration of thymidine. To monitor how the labeled thymidine is processed in the body, investigators will analyze urine from the child's diapers. Each time a diaper is changed, a cotton ball will be placed in the diaper. At the next diaper change, this cotton ball will be removed from the diaper, placed in a Ziploc bag, and stored in the freezer. They will be collected and stored cotton balls starting with the first administration of thymidine until 24 hours after the last administration. The frozen cotton balls may be collected from the home by a nurse or brought by parent to the next clinic visit.
Procedure: Echocardiogram — On Study Day 1 to obtain baseline assessment of cardiac size. A second research dedicated echocardiogram will be done after being anesthetized for surgery. Echocardiography is routinely performed to determine right ventricle (RV) structure of the heart and function in Tetrology of Fallot/ Pulmonary Stenosis (ToF/PS) and is non-invasive.
Procedure: Cardiac MRI (CMR) — A limited study protocol will be performed using the feed-and-bundle technique at the time of study enrollment, The feed and bundle technique is utilized so that the infant will be as comfortable as possible and asleep during the procedure. This is done to prevent the risk of sedation and allow for a more natural sleep. The baby is undressed, prepared with ECG-leads and an oxygen saturation probe, and fed. With this "feed, swaddle, and sleep" technique, scanning times of 30-60 minutes can be achieved, which provides the stillness needed for accurate visualization of the heart. A second CMR, with the same limited study protocol, will be performed under general anesthesia prior to surgical repair. It does not pose any risk of radiation exposure and will not require IV placement or contrast administration for a limited assessement of the right ventricle.
Drug: Propranolol Hydrochloride — For patients who are randomized to receive propranolol, The target dose for this study will be 4 mg/kg/day divided in 4 doses. The first dose will be given in the Pediatric Clinical and Translational Research Center (PCTRC) at 1mg/kg. Parents will administer propranolol (1 mg/kg po x 4 doses per day). Parents will be instructed to administer propranolol with feeding or soon after feeding, but not before feeding. families will also be given instructions for regarding 15N-thymidine dosing frequency and interval and provided with a log sheet to record administered and missed doses of propranolol and 15N-thymidine.
  Other Names: Propranolol
  Arms: Propranolol
Drug: Placebo — For patients who are randomized to receive placebo, the first dose will be given in the Pediatric Translational Research Center (PCTRC) and will be based on the patients weight. Parents will administer placebo 4 doses per day. Treatment with placebo will begin at 1 month of age and continue until 4 months of age or 24hrs prior to surgical repair, whichever comes first.
  Arms: Placebo
Procedure: Physical Exam — On Study Day 1; monthly until surgery in conjunction with patient's clinical cardiology appointment; and at the time of surgery. Will include vital signs.
Other: Specimen Collection — On the morning of surgery, after IV access is obtained for anesthesia 2 ml of blood will be collected for analysis. A small piece of heart tissue and fat that has already been removed during surgery will be collected for analysis.

SUMMARY:
Heart failure is a common long-term complication in patients with congenital heart disease (CHD). Medical treatments to promote regeneration of new healthy heart muscle cells have the potential to provide new heart failure treatments for these patients. The development of such therapies is limited by the poor understanding of the ways in which heart muscles grow after birth. Investigators have learned that humans without heart disease generate new heart muscles cells up to the age of 20 years old and that this is decreased in patients with congenital heart disease like Tetralogy of Fallot. Investigators are trying to determine if treatment with a medicine called Propranolol can increase heart muscle cell proliferation and, with that, normalize heart growth. Investigators will examine discarded heart muscle tissue that is obtained during surgery for the presence of new heart muscle cells. Propranolol is approved by the Food and Drug Administration (FDA) to treat a certain kind of benign tumor in infants (hemangioma), but it is not currently approved by the FDA to increase heart muscle growth.

ELIGIBILITY:
Inclusion Criteria:

* Male and female infants < 60 days of age with a diagnosis of tetralogy of Fallot (ToF) with pulmonary stenosis (PS) or double outlet right ventricle (DORV), tetralogy type by echocardiogram, who weigh greater than 2 kg at the time of consent and are tolerating enteral feeds.
* DORV variant

Exclusion Criteria:

* congenital atrio-ventricular block on EKG (PR interval > 120 ms),
* concomitant medication administration that interacts with propranolol,
* patient family is, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason,
* gestation age < 35 weeks,
* infants of diabetic mothers, asthma or underlying respiratory disease,
* presence of metal implants in infants.

Ages: 30 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiomyocyte Division | At the time of complete surgical repair, at approximately 3-9 months old, it is expected that a piece of RV myocardium will be resected. This tissue will be collected and analyzed using a multiple isotope mass spectrometer.
  To quantify cardiomyocyte division, investigators will utilize previously established MIMS (membrane introduction mass spectrometry) approach. Briefly, investigators will administer 5 enteral doses of 15N-thymidine to all patients at 1 month after birth. Cardiomyocytes that have undergone DNA replication after the intake of 15N-thymidine will incorporate the stable isotope into their DNA.

SECONDARY OUTCOMES:
Hypertrophy as assessed by echocardiography | At 1 month and at time of surgery
  Analysis of the impact of propranolol on Right Ventricle Myocardial Volume
Hypertrophy as assessed by Cardiac MRI | At 1 month and at time of surgery
  Analysis of the impact of propranolol on Right Ventricle Myocardial Volume
Hypertrophy assessed by microscopy | At time of Surgery
  Analysis of the impact of propranolol on cardiomyocytes cross sectional area

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Kuhn, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Weill Cornell Medicine, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Upmc Children'S Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Khoudary SR, Fabio A, Yester JW, Steinhauser ML, Christopher AB, Gyngard F, Adams PS, Morell VO, Viegas M, Da Silva JP, Da Silva LF, Castro-Medina M, McCormick A, Reyes-Mugica M, Barlas M, Liu H, Thomas D, Ammanamanchi N, Sada R, Cuda M, Hartigan E, Groscost DK, Kuhn B. Design and rationale of a clinical trial to increase cardiomyocyte division in infants with tetralogy of Fallot. Int J Cardiol. 2021 Sep 15;339:36-42. doi: 10.1016/j.ijcard.2021.07.020. Epub 2021 Jul 12. PMID 34265312